CLINICAL TRIAL: NCT03852394
Title: Influence of Respiratory Mechanics on Diaphragmatic Dysfunction in COPD Patients Who Have Failed Non-invasive Mechanical Ventilation
Brief Title: Influence of Respiratory Mechanics on Diaphragmatic Dysfunction in COPD Patients Who Have Failed NIV (RHYDIAN)
Acronym: RHYDIAN
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Alessandro Marchioni, Principal Investigator, University of Modena and Reggio Emilia
Other Study IDs: UModenaReggio 4
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Diaphragm Dysfunction; COPD Exacerbation; Mechanical Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Respiratory mechanics assessment — The study protocol consisted of two consecutive phases; in the first step measurements of static respiratory mechanics and end expiratory lung volume (EELV) were performed after 30 minutes of MV in volume control mode. In the second step transdiaphragmatic pressure (Pdi) was calculated by means of a sniff maneuver (Maximal Pdi) after 30 minutes of spontaneous breathing trial. Linear regression analysis and Pearson's correlation coefficient was used to asses the association between Maximal Pdi values and static and dynamic mechanical features and the association between Maximal Pdi and Pdi/Maximal Pdi.

SUMMARY:
Although non-invasive mechanical ventilation (NIV) is the gold standard treatment for patients with acute exacerbation of COPD (AECOPD) who develop respiratory acidosis, failure rate are still high ranging from 5% to 40%. Recent studies have shown that the onset of severe diaphragmatic dysfunction (DD) during AECOPD increases risk of NIV failure and mortality in this subset of patients. Although the imbalance between the load and the contractile capacity of inspiratory muscles seems the main cause of AECOPD-induced hypercapnic respiratory failure, data regarding the influence of mechanical derangement on diaphragmatic performance in this acute phase are lacking. With this study we aim at investigating the impact of respiratory mechanics on diaphragm function in AECOPD patients who experienced NIV failure. AECOPD with respiratory acidosis admitted to the ICU of the University Hospital of Modena from 2017-2018 undergoing mechanical ventilation (MV) due to NIV failure were enrolled. The study protocol consisted of two consecutive phases; in the first step measurements of static respiratory mechanics and end expiratory lung volume (EELV) were performed after 30 minutes of MV in volume control mode. In the second step transdiaphragmatic pressure (Pdi) was calculated by means of a sniff maneuver (Maximal Pdi) after 30 minutes of spontaneous breathing trial. Linear regression analysis and Pearson's correlation coefficient was used to asses the association between Maximal Pdi values and static and dynamic mechanical features and the association between Maximal Pdi and Pdi/Maximal Pdi.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years
* AECOPD with respiratory acidosis admitted to the Respiratory Intensive Care Unit of the University Hospital of Modena (Italy) undergoing endotracheal intubation due to NIV failure.

Exclusion Criteria:

* history of neuromuscular disease,
* presence of chest wall deformities,
* coexistence of interstitial lung disease,
* presence of pulmonary edema,
* severe hemodynamic instability,
* septic shock,
* evidence of lobar pneumonia or bilateral parenchymal consolidation at chest X-ray on admission,
* contraindication to NIV,
* previously assessed diaphragmatic palsy,
* intracranial hypertension,
* known pregnancy,
* need for immediate endotracheal intubation,
* neurologic impairment,
* lack of collaboration,
* unreliable maneuver to calculate maximal transdiaphragmatic pressure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort study
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Impact of static elastance on diaphragm function in AECOPD patient who failed NIV | 30 days from Respiratory Intensive Care Unit admission
  Correlation between static elastance and Maximal Pdi in patients undergoing mechanical ventilation for AECOPD
Impact of dynamic intrinsic Positive End Expiratory Pressure on diaphragm function in AECOPD patient who failed NIV | 30 days from Respiratory Intensive Care Unit admission
  Correlation between dynamic intrinsic Positive End Expiratory Pressure and Maximal Pdi in patients undergoing mechanical ventilation for AECOPD

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Modena Policlinico di Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Undecided